## Cover Page for ClinicalTrials.gov

**Document: Informed Consent Form** 

Title: Efficacy Of Pyodine Soaked Gelfoam Vs Single Topical Application Of Clotrimazole In Treatment Of Otomycosis: A Randomized

Controlled Clinical Trial

**Document Date: 16-June-2023** 

Zuneera Shabbir

## **CONSENT FORM**

## Department of Rawalpindi Medical University and Allied Hospitals, RAWALPINDI

Title of the study: Efficacy Of Pyodine Soaked Gelfoam Vs Single Topical Application Of Clotrimazole In Treatment Of Otomycosis: A Randomized Controlled Clinical Trial By Dr. Zuneera Shabbir

| Name: |
|---|
| Guardian's name/relation: |
| Hospital A&D No: |
| • I confirm that I have read and understood the information about the project as provided in the Participant Information Sheet dated [Insert Date]. |
| <ul> <li>I confirm that I have had the opportunity to ask questions and the researcher has<br/>answered any questions about the study to my satisfaction.</li> </ul> |
| • I understand that my participation is voluntary and that I am free to withdraw from the project at any time, without having to give a reason and without any consequences. |
| • I understand that I can withdraw my data from the study at any time. |
| • I understand that any information recorded in the investigation will remain confidential and no information that identifies me will be made publicly available. |
| • I consent use of this data in research, publications, sharing and archiving as explained in the Participant Information Sheet. |
| <ul> <li>I consent for audio/ video/ interviews recordings as part of the project Yes/ No</li> <li>I agree / do not agree (delete as appropriate) to take part in the above study.</li> </ul> |
| Name of Participant Date / Guardians Signature: |
| Doctor: Zuneera Shabbir |
| Date / Signature |

Interview Signature Date: